CLINICAL TRIAL: NCT02311140
Title: Effects of Kalydeco on Upper Airway and Paranasal Sinus Inflammation Measured by Nasal Lavage and on Symptoms
Acronym: KPNSI
Status: Completed | Type: Observational
Sponsor: University of Jena (Other)
Collaborators: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Prof. Dr. Jochen G. Mainz, Head of CF Center, Pediatric Pulmonology, University of Jena
Other Study IDs: UKJ-IVA-Nasal
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Inflammatory Changes in Epithelial Lining Fluid Sampled Non-invasively by Nasal Lavage in CF Patients With G551D Receiving Kalydeco
Keywords: cystic fibrosis; nasal lavage; inflammation; Interleukin (IL)-6; IL-8; pulmonary function
MeSH Terms: conditions — Cystic Fibrosis; Inflammation | interventions — Nasal Lavage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasal lavage
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cystic Fibrosis patients with G551D mutation: Cohort Description Ten participants (6 Jena/4 Innsbruck) were included, of whom 6 were female and 4 were male. At the start of the study, patients were aged 7-45 years (mean age: 16.55 ± 13.42 years). Results of sweat tests and lung function FEV1 were available only from 8 patients. Lung function at baseline, as obtained from those patients, ranged from 0.96 to 4.07 L (mean FEV1: 99.7 ± 20.3% predicted, median: 103.6% predicted, IQR=20.4% predicted).
  Interventions: Other: nasal lavage (routine diagnostic procedure in our centre), assessment of symptoms

INTERVENTIONS:
Other: nasal lavage (routine diagnostic procedure in our centre), assessment of symptoms

SUMMARY:
The aim of the proposed trial in assessment of effects of Kalydeco™ treatment on sinonasal involvement in CF patients with at least one mutation of G551D receiving a new therapy with the CFTR potentiator. The focus will be given on changes in epithelial lining fluid inflammatory markers from CF upper airways sampled by nasal lavage.

The program is subdivided into a part A assessing inflammatory markers in NL and sinonasal symptoms longitudinally from pre-treatment to months with the new therapy.

Part B will only be performed in a smaller subgroup and assess inflammatory markers in NL every second day in the first month of treatment and then every week until the end of month 3 with Kalydeco™ therapy.

DETAILED DESCRIPTION:
Enrollment of Patients In this longitudinal trial, 10 CF patients with a G551D mutation, newly receiving ivacaftor 150 mg bid, as approved (1), were included in the Jena (Germany) and Innsbruck (Austria) University CF centers. Inclusion criteria were: CF patients' age ≥ 6 years with a diagnosis confirmed by two positive sweat tests and/or detection of two disease-causing CFTR mutations; one of them being G551D. Patients were required to strictly follow the procedures defined in the SOPs and they and/or their parents gave informed written consent prior to enrolment. Exclusion criteria were: inability to perform NL in a standardized manner as described below, contraindication for ivacaftor, pregnancy or breast-feeding, and participation in another clinical study within 30 days prior to study drug administration. Nasal Lavage Patients were thoroughly trained to perform NL in standardized home-based conditions (Figures 1A-C) by using the instructionvideo from our publication in Journal of Immunological Methods 2014 (14) and an illustrated SOP sheet. The pooled native NLF was transferred into disposed reaction tubes containing 15 μL of protease inhibitor (Figures 1D, E) and, within 30 minutes after sampling, stored in a freezer below -18°C until transfer on ice to the centers. Here, the vials were directly stored at - 80°C until performance of laboratory analyses. Prior to the initiation of ivacaftor therapy, NL was collected at least once a week (mean: 5.5 ± 3.9 samplings/patient) during a mean time of 30.3 ± 19.7 days. During the first month of therapy (days 0-30), NL was collected every second day and once/week from month two onward (mean: 25.9 ± 4.1 samplings/patient). Follow-up range after initiation of ivacaftor: 2.3-16.1 months, (median: 5.7 months). Assessment of Inflammatory Mediators Concentrations of IL-1b, IL-6, and IL-8 were measured in undiluted NL fluid using Milliplex® MAP Kits (Human High Sensitivity HS TCMAG-28K, Merck Millipore; Darmstadt, Germany) and a Bio-Plex® 200 system (Bio-Rad; Hercules, California, USA) according to the manufacturer's instructions. Measurements of Neutrophil Elastase (NE) were performed using Human PMN Elastase ELISA (DEH3311, Demeditec Diagnostics GmbH; Kiel, Germany) and read by a FLUOstar Galaxy spectrometer (BMG LABTECH GmbH; Offenburg, Germany). As specified by the manufacturer, lower detection limits were 0.12 pg/mL (IL-1b), 0.13 pg/mL (IL-6), 0.12 pg/mL (IL-8), and 0.2 ng/mL (NE). Statistical Analyses Descriptive statistics were used to describe clinical characteristics of the study population. Linear mixed-effects models were performed to analyze overall trends of inflammatory markers. To smooth effects caused by outliers in inflammatory marker values, individual changes regarding cumulative periods for each patient were determined by calculating medians for the time periods before and after treatment initiation (i.e. regarding periods of 4, 8 and 12 weeks during treatment as shown in Figure 2). The resulting individual patients' medians were used to calculate medians and interquartile ranges (IQR) of the entire cohort at the end of the above-mentioned time periods. Wilcoxon signedrank test (two-tailed) was applied to determine changes in the aforementioned inflammatory mediators, sweat test, FEV1 and their statistical significance (using p<0.05) during the new therapy. All statistical analyses were performed with IBM SPSS 19 (SPSS Inc., Chicago, IL, USA); figures were created with GraphPad Prism (GraphPad Software Inc., La Jolla, CA, USA).

ELIGIBILITY:
Inclusion Criteria:

* G551D and Kalydeco therapy

Exclusion Criteria:

* no G551D

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CF patients with G551D mutation receiving Kalydeco
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-07; Primary Completion 2017-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Changes in concentration of inflammatory markers | 3 yrs
  Concentrations of IL-1b, IL-6, and IL-8 were measured in undiluted NL fluid using Milliplex® MAP Kits (Human High Sensitivity HS TCMAG-28K, Merck Millipore; Darmstadt, Germany) and a Bio-Plex® 200 system (Bio-Rad; Hercules, California, USA) according to the manufacturer's instructions. Measurements of Neutrophil Elastase (NE) were performed using Human PMN Elastase ELISA (DEH3311, Demeditec Diagnostics GmbH; Kiel, Germany) and read by a FLUOstar Galaxy spectrometer (BMG LABTECH GmbH; Offenburg, Germany). As specified by the manufacturer, lower detection limits were 0.12 pg/mL (IL-1b), 0.13 pg/mL (IL-6), 0.12 pg/mL (IL-8), and 0.2 ng/mL (NE).

CONTACTS AND LOCATIONS:
Locations (1):
- Jena University Hospital, CF Center, Jena, Germany

REFERENCES:
- [Result] Mainz JG, Arnold C, Wittstock K, Hipler UC, Lehmann T, Zagoya C, Duckstein F, Ellemunter H, Hentschel J. Ivacaftor Reduces Inflammatory Mediators in Upper Airway Lining Fluid From Cystic Fibrosis Patients With a G551D Mutation: Serial Non-Invasive Home-Based Collection of Upper Airway Lining Fluid. Front Immunol. 2021 May 5;12:642180. doi: 10.3389/fimmu.2021.642180. eCollection 2021. PMID 34025651